CLINICAL TRIAL: NCT06980506
Title: Imaging of Patients With Solid Tumor Cancer Via Intermediate-Size Patient Population Expanded Access Investigational New Drug (IND)
Brief Title: MNPR-101-DFO*-89Zr Expanded Access Program (EAP) for Patients With Solid Tumor Cancer
Status: Available | Type: Expanded Access
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IST-00Ca
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Solid Tumor; Solid Tumor, Adult
Keywords: Solid Tumor; PET/CT; urokinase plasminogen activator receptor; uPAR; Zirconium-89 imaging; Positron emission tomography/computed tomography; MNPR-101-DFO*-89Zr; uPAR-positive; Urokinase plasminogen activator receptor-positive; EAP IST-00Cb; Antibody radionuclide conjugate; Monoclonal antibody radionuclide conjugate; Solid tumor imaging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Diagnostic Test: MNPR-101-DFO*-89Zr — MNPR-101-DFO*-89Zr is an antibody radionuclide conjugate intended to image solid tumors expressing uPAR.

SUMMARY:
The purpose of this Expanded Access Program (EAP) is to allow use of the investigational imaging agent, MNPR-101-DFO*-89Zr, with positron emission tomography/computed tomography (PET/CT) imaging, to non-invasively detect the presence of urokinase plasminogen activator receptor (uPAR) binding in solid tumors. uPAR binding is higher in tumors compared to normal tissue in some cancers.

DETAILED DESCRIPTION:
Imaging agent MNPR-101-DFO*-89Zr will be dosed to adult patients diagnosed with solid tumor cancer followed 3 to 5 days later by PET/CT imaging. The result will determine if there is sufficient uPAR binding, as assessed by the Investigator, to support administration of the companion intervention MNPR-101-PCTA-177Lu in a separate expanded access program (EAP IST-00Cb). The safety of MNPR-101-DFO*-89Zr will be evaluated as will the amount of radioactivity present in blood samples.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor cancer that is refractory to existing therapy(ies) known to provide clinical benefit, or for which no standard treatment is available, or is contraindicated
* Ability to understand and willingness to sign a written informed consent document

Key Exclusion Criteria:

* Continuing ≥ Grade 3 adverse reactions from prior systemic therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0)
* Prior treatment with any radiopharmaceutical or investigational agents within 4 weeks or 5 half-lives, whichever is longer, prior to administration of MNPR-101-DFO*-89Zr
* Evidence of impaired organ function, particularly bone marrow, liver, kidney, or heart, according to specific test parameters
* Presence of other serious, non-malignant diseases or any other condition that, in the opinion of the investigator, could interfere with the objectives of the study, participant safety, or compliance.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S. Delpassand, M.D. Chairman & Medical Director, Nuclear Medicine, Principal Investigator — Excel Diagnostics & Nuclear Oncology Center
Locations (1):
- Excel Diagnostics & Nuclear Oncology Center, Houston, Texas, United States